CLINICAL TRIAL: NCT05901389
Title: Effects of Continuous Lidocaine Infusion Via Closed Chest Drainage Tube on Postoperative Analgesia for Patients Undergoing Thoracoscopic Partial Lung Resection: a Single-center Randomized Controlled Clinical Trial
Brief Title: Continuous Lidocaine Infusion Via Closed Chest Drainage Tube for Pain Control After Thoracoscopic Partial Lung Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KYLL-202210-071-1
Record Dates: First submitted 2023-05-03; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-01

CONDITIONS: Lidocaine; Analgesia; Pain, Postoperative; Thoracic Surgery
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: lidocaine will be injection by electronic analgesic pump, and the pulse infusion speed is 1ml / 30min, and 2ml / h for continuous infusion
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lidocaine (Experimental): Patients in this group will receive continuous lidocaine infusion via closed chest drainage tube. The pulse infusion speed is 1ml / 30min, and the continuous infusion speed was 2ml / h.
  Interventions: Drug: Lidocaine
- normal saline (Placebo Comparator): Patients in this group will receive continuous normal saline infusion via closed chest drainage tube. The pulse infusion speed is same as the lidocaine group.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Lidocaine — After the thoracoscopic surgery, lidocaine will be transfused through the epidural tube fixed in the chest drainage tube was connected to an electronic pump whose parameters are already set up (marking the chest drain for analgesia).
  Arms: lidocaine
Drug: normal saline — After the thoracoscopic surgery, normal saline will be transfused through the epidural tube fixed in the chest drainage tube was connected to an electronic pump whose parameters are already set up (marking the chest drain for analgesia).
  Arms: normal saline

SUMMARY:
The goal of this clinical trial is to learn about the effects on postoperative analgesia of continuous lidocaine infusion via closed chest drainage tube for patients undergoing thoracoscopic partial lung resection. The main questions it aims to answer are:

* To explore whether continuous lidocaine pumping via closed chest drainage tube has good analgesic and anti-inflammatory effects for patients undergoing partial thoracoscopic pneumonectomy.
* Whether the multimodal analgesia combined with continuous lidocaine pump can reduce the postoperative application of opioids, reduce the occurrence of postoperative complications, and promote the recovery of postoperative lung function and accelerate recovery.

For participants who undergoing the thoracoscopic partial lung resection with postoperative indwelling drainage tube, the epidural tube fixed in the drainage tube is connected to the completed infusion pump (marking the chest drain for analgesia). The comparison group only accept the intravenous analgesia after surgery.

DETAILED DESCRIPTION:
At present, multimodal analgesia has been the most commonly used approaches for the treatment of postoperative pain of thoracic surgery, including steroidal anti-inflammatory drugs, administration of opioid, and local anesthesia.

The investigators found that continuous lidocaine analgesia with local anesthesia through thoracic closed drainage tube could improve postoperative pain caused by drainage tube retention, reduce postoperative pain score, and improve postoperative recovery of respiratory function in patients. In the protocol, lidocaine was continuously pumped with a superficial anesthetic effect on the pleura, while mucosal absorption was almost equivalent to intravenous infusion, so its systemic anti-inflammatory effect is also explored.

In the protocol，participants will be randomized in a 1:1 ratio to the control or experimental groups. The experimental group received a continuous infusion of lidocaineThe experimental group used 2% lidocaine 100ml, and the control group was the conventional treatment group. The control group received only standard intravenous analgesia。In addition to receiving simple intravenous analgesia, the experimental group also received continuous infusion of lidocaine in the pleural cavity.

ELIGIBILITY:
Inclusion Criteria:

1. participants ages 18-70 years.
2. participants undergoing thoracoscopic partial lung resection with an indwelling drainage tube after surgery.
3. American Society of Anesthesiologists classification (ASA)I-III.

Exclusion Criteria:

1. severe heart failure, cardiac arrhythmias,the New York Heart Association(NYHA) classification≥III.
2. hypersensitivity to lidocaine,History of local anesthetic poisoning.
3. severe renal or hepatic dysfunction.
4. body mass index (BMI)>35 kg m-2.
5. severe pleural adhesions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
postoperative pain score（NRS） | Day 1
  The full name of NRS score is Numerical Rating Scale. The minimum value of NRS score is 0 and the maximum value is 10. Patients can score themselves according to the pain level corresponding to the number, A score of 0 represents painless, 1-3 represents mild pain, 4-6 represents moderate pain and should be intervened, 7-10 represents severe pain and requires urgent treatment. In this study,the investigators mainly investigated the incidence of postoperative pain score was greater than 3 in each group.

SECONDARY OUTCOMES:
Changes in postoperative pain | Day 2
  Changes in postoperative pain score (NRS) at 12h and 48h until extubation. The full name of NRS score is Numerical Rating Scale. The minimum value of NRS score is 0 and the maximum value is 10. Patients can score themselves according to the pain level corresponding to the number, A score of 0 represents painless, 1-3 represents mild pain, 4-6 represents moderate pain and should be intervened, 7-10 represents severe pain and requires urgent treatment.
the use of flurbiprofen axetil | Day 3
  the amount of rescue analgesic drugs flurbiprofen axetil used
the use of dolantin | Day 3
  the amount of rescue analgesic drugs dolantin used
the use of opioids | Day 2
  total amount of opioid use within 48h after surgery
postoperative adverse events | Day 3
  the incidence of nausea, vomiting, and vertigo after surgery
the amount of postoperative wound drainage | Day 3
  total amount of fluid drained after surgery
C-reactive protein | Day 1
  The inflammatory marker of participants will be test after surgery
interleukin-6 | Day 1
  The inflammatory marker of participants will be test after surgery
postoperative delusion | Day 3
  The incidence of postoperative delusion.
drainage extraction | up to 24 hours (before extubation)
  The time taken for the patient to remove the drain after surgery
ICU stay time | From date of ICU admission until the date of leaving ICU, assessed up to 5 days.
  The length of time the patient remains in the ICU.
postoperative pulmonary complications | Day 3
  The probability of patients acquiring pulmonary complications after surgery.
hospital length of stay | From date of hospital admission until the date of discharge,assessed up to 15 days.
  The time between hospital admission and discharge
healing rate of drainage wound | Day 21
  The healing rate of drainage wound at 21 days after surgery.
readmission rate | Month 1
  The readmission rate of patients in one month after surgery.

REFERENCES:
- [Background] Abdallah FW, Brull R. Is sciatic nerve block advantageous when combined with femoral nerve block for postoperative analgesia following total knee arthroplasty? A systematic review. Reg Anesth Pain Med. 2011 Sep-Oct;36(5):493-8. doi: 10.1097/AAP.0b013e318228d5d4. PMID 21857266
- [Background] Barletta M, Reed R. Local Anesthetics: Pharmacology and Special Preparations. Vet Clin North Am Small Anim Pract. 2019 Nov;49(6):1109-1125. doi: 10.1016/j.cvsm.2019.07.004. Epub 2019 Aug 30. PMID 31474415
- [Background] Becker DE, Reed KL. Local anesthetics: review of pharmacological considerations. Anesth Prog. 2012 Summer;59(2):90-101; quiz 102-3. doi: 10.2344/0003-3006-59.2.90. PMID 22822998
- [Background] Camorcia M, Capogna G, Columb MO. Effect of sex and pregnancy on the potency of intrathecal bupivacaine: determination of ED(5)(0) for motor block with the up-down sequential allocation method. Eur J Anaesthesiol. 2011 Apr;28(4):240-4. PMID 21513074
- [Background] Capdevila X, Pirat P, Bringuier S, Gaertner E, Singelyn F, Bernard N, Choquet O, Bouaziz H, Bonnet F; French Study Group on Continuous Peripheral Nerve Blocks. Continuous peripheral nerve blocks in hospital wards after orthopedic surgery: a multicenter prospective analysis of the quality of postoperative analgesia and complications in 1,416 patients. Anesthesiology. 2005 Nov;103(5):1035-45. doi: 10.1097/00000542-200511000-00018. PMID 16249678
- [Background] Choquet O, Noble GB, Abbal B, Morau D, Bringuier S, Capdevila X. Subparaneural versus circumferential extraneural injection at the bifurcation level in ultrasound-guided popliteal sciatic nerve blocks: a prospective, randomized, double-blind study. Reg Anesth Pain Med. 2014 Jul-Aug;39(4):306-11. doi: 10.1097/AAP.0000000000000095. PMID 24918330
- [Background] Dalkilic N, Tuncer S, Burat I. Dexmedetomidine augments the effect of lidocaine: power spectrum and nerve conduction velocity distribution study. BMC Anesthesiol. 2015 Mar 6;15:24. doi: 10.1186/s12871-015-0009-9. eCollection 2015. PMID 25762864
- [Background] De Buck F, Devroe S, Missant C, Van de Velde M. Regional anesthesia outside the operating room: indications and techniques. Curr Opin Anaesthesiol. 2012 Aug;25(4):501-7. doi: 10.1097/ACO.0b013e3283556f58. PMID 22673788
- [Background] Desmet M, Braems H, Reynvoet M, Plasschaert S, Van Cauwelaert J, Pottel H, Carlier S, Missant C, Van de Velde M. I.V. and perineural dexamethasone are equivalent in increasing the analgesic duration of a single-shot interscalene block with ropivacaine for shoulder surgery: a prospective, randomized, placebo-controlled study. Br J Anaesth. 2013 Sep;111(3):445-52. doi: 10.1093/bja/aet109. Epub 2013 Apr 15. PMID 23587875
- [Background] Drachman D, Strichartz G. Potassium channel blockers potentiate impulse inhibition by local anesthetics. Anesthesiology. 1991 Dec;75(6):1051-61. doi: 10.1097/00000542-199112000-00018. PMID 1741497
- [Background] Durham SD, Flournoy N, Rosenberger WF. A random walk rule for phase I clinical trials. Biometrics. 1997 Jun;53(2):745-60. PMID 9192462
- [Background] Elmas C, Atanassoff PG. Combined inguinal paravascular (3-in-1) and sciatic nerve blocks for lower limb surgery. Reg Anesth. 1993 Mar-Apr;18(2):88-92. PMID 8489988
- [Background] Grape S, Kirkham KR, Baeriswyl M, Albrecht E. The analgesic efficacy of sciatic nerve block in addition to femoral nerve block in patients undergoing total knee arthroplasty: a systematic review and meta-analysis. Anaesthesia. 2016 Oct;71(10):1198-209. doi: 10.1111/anae.13568. Epub 2016 Jul 29. PMID 27469381
- [Background] Green SB. How Many Subjects Does It Take To Do A Regression Analysis. Multivariate Behav Res. 1991 Jul 1;26(3):499-510. doi: 10.1207/s15327906mbr2603_7. PMID 26776715
- [Background] Gupta PK, Pace NL, Hopkins PM. Effect of body mass index on the ED50 volume of bupivacaine 0.5% for supraclavicular brachial plexus block. Br J Anaesth. 2010 Apr;104(4):490-5. doi: 10.1093/bja/aeq017. Epub 2010 Feb 18. PMID 20167584
- [Background] He M, Ling DD, Cai GY, Zou TX, Yu B. Two different placement paths in popliteal fossa with a novel nerve block needle for postoperative analgesia after foot and ankle surgery. Minerva Anestesiol. 2018 May;84(5):582-589. doi: 10.23736/S0375-9393.17.12061-4. Epub 2017 Oct 12. PMID 29027771
- [Background] Kang R, Jeong JS, Yoo JC, Lee JH, Choi SJ, Gwak MS, Hahm TS, Huh J, Ko JS. Effective Dose of Intravenous Dexmedetomidine to Prolong the Analgesic Duration of Interscalene Brachial Plexus Block: A Single-Center, Prospective, Double-Blind, Randomized Controlled Trial. Reg Anesth Pain Med. 2018 Jul;43(5):488-495. doi: 10.1097/AAP.0000000000000773. PMID 29630034
- [Background] Keplinger M, Marhofer P, Marhofer D, Schroegendorfer K, Haslik W, Zeitlinger M, Mayer CV, Kettner SC. Effective local anaesthetic volumes for sciatic nerve blockade: a clinical evaluation of the ED99. Anaesthesia. 2015 May;70(5):585-90. doi: 10.1111/anae.13013. Epub 2015 Jan 20. PMID 25644578
- [Background] Kettner SC, Willschke H, Marhofer P. Does regional anaesthesia really improve outcome? Br J Anaesth. 2011 Dec;107 Suppl 1:i90-5. doi: 10.1093/bja/aer340. PMID 22156274
- [Background] Latzke D, Marhofer P, Zeitlinger M, Machata A, Neumann F, Lackner E, Kettner SC. Minimal local anaesthetic volumes for sciatic nerve block: evaluation of ED 99 in volunteers. Br J Anaesth. 2010 Feb;104(2):239-44. doi: 10.1093/bja/aep368. Epub 2009 Dec 23. PMID 20034967
- [Background] Lirk P, Hollmann MW, Strichartz G. The Science of Local Anesthesia: Basic Research, Clinical Application, and Future Directions. Anesth Analg. 2018 Apr;126(4):1381-1392. doi: 10.1213/ANE.0000000000002665. PMID 29189280
- [Background] Marhofer P, Pilz-Lubsczyk B, Lonnqvist PA, Fleischmann E. Ultrasound-guided peripheral regional anaesthesia: a feasibility study in obese versus normal-weight women. Int J Obes (Lond). 2014 Mar;38(3):451-5. doi: 10.1038/ijo.2013.119. Epub 2013 Jun 25. PMID 23797187
- [Background] Nathan N, Benrhaiem M, Lotfi H, Debord J, Rigaud G, Lachatre G, Adenis JP, Feiss P. The role of hyaluronidase on lidocaine and bupivacaine pharmacokinetics after peribulbar blockade. Anesth Analg. 1996 May;82(5):1060-4. doi: 10.1097/00000539-199605000-00032. PMID 8610868
- [Background] O'Donnell BD, Iohom G. An estimation of the minimum effective anesthetic volume of 2% lidocaine in ultrasound-guided axillary brachial plexus block. Anesthesiology. 2009 Jul;111(1):25-9. doi: 10.1097/ALN.0b013e3181a915c7. PMID 19512869
- [Background] Palmer CG, Jagannathan S. Sciatic nerve block and enhanced recovery after total knee arthroplasty. Anaesthesia. 2016 Dec;71(12):1495. doi: 10.1111/anae.13728. No abstract available. PMID 27870171
- [Background] Raymond SA, Steffensen SC, Gugino LD, Strichartz GR. The role of length of nerve exposed to local anesthetics in impulse blocking action. Anesth Analg. 1989 May;68(5):563-70. PMID 2785778